CLINICAL TRIAL: NCT04610190
Title: Useability Test of Gait Enhancing and Motivating System-Hip (GEMS-H)
Brief Title: Useability Test to the Wearable Walking-assist Robot (GEMS-H) for Normal Adults Including the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yun-Hee Kim (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Sponsor-Investigator, Yun-Hee Kim, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-10-016
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Gait Disorders in Old Age
Keywords: Wearable hip assist robot; Gait; User test; Robot gait training; Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training with Gait Enhancing and Motivating System (GEMS-H) Robot (Experimental): Training consists of 15 minutes task-specific training and 20-30 minutes functional gait training on varied environments with device.
  Interventions: Device: Training with Gait Enhancing and Motivating System (GEMS-H) Robot

INTERVENTIONS:
Device: Training with Gait Enhancing and Motivating System (GEMS-H) Robot — Training consists of 15 minutes task-specific training and 30 minutes functional gait training on varied environments with device.
  Other Names: Training with GEMS-H

SUMMARY:
The purpose of this study is to investigate the userbility and satisfaction of functional gait training with the Gait Enhancing and Motivating System-Hip type (GEMS-H) on locomotor function in normal adults including the elderly.

DETAILED DESCRIPTION:
The GEMS-H is a hip-type assist device developed by the Samsung Advanced Institute of Technology. The GEMS-H is worn around the waist and fastened at the waist and thighs by a set of belts with velcro to assist motion at the hip joints. The device weighs 2.1kg, and has 2 brushless direct current motors running on a rechargeable lithium ion battery. The normal operation time for the device is 2 hours. The GEMS-H is available in three sizes to fit various waist/hip sizes: small, medium, and large. The width of each version can be adjusted further to fit individual body size within the circumference range. Also, the thigh frames are available in three sizes (large, medium, and small) for different leg lengths. It is controlled through a custom built application on a hand held tablet.

Participants will be normal adults with community-dwelling older adults aged 19-85.

Participants will be scheduled for 24 training sessions of training plus 3 sessions of testing (pre-training, mid-test after the 12 sessions of training, post-training).

ELIGIBILITY:
Inclusion Criteria:

* Age: 19 - 85 years
* Living in the community-dwelling with ability to travel to the intervention site to participate in the training program.

Exclusion Criteria:

* Difficult to understand experimental tasks because of extremely severe cognitive impairment (Korean-Mini-Mental State Examination, K-MMSE≤10)
* Serious cardiac conditions (hospitalization for myocardial infarction or heart surgery within 3 months, history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living)
* BMI ≥ 35 kg/m2
* Serious medical conditions including myocardial infarction or heart surgery within 3 months, history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living, Severe hypertension, severe weight bearing pain, life expectancy less than one year

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in 10 meter walk test from baseline in gait speed | session 0 (initial visit); after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  Measure of self selected speeds by measuring the time it takes an individual to walk 10 meters. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."

SECONDARY OUTCOMES:
Change in Berg Balance Scale (BBS) from baseline in balance | session 0 (initial visit); after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  Measure of balance function. A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Score the LOWEST performance. Total Score = 56.
Change in Timed Up and Go test (TUG) from baseline in balance | session 0 (initial visit); after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  Measure of dynamic balance function. 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention. A score of 30 seconds or more suggests that the person may be prone to falls.
Changes in Functional Reach Test (FRT) from baseline | session 0 (initial visit); after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  FRT is a single item test developed as a quick screen for balance problems. Measurement Interpretation: 10"/25 cm or greater Low risk of falls; 6"/15cm to 10"/25cm Risk of falling is 2x greater than normal; 6"/15cm or less Risk of falling is 4x greater than normal; Unwilling to reach Risk of falling is 8x greater than normal.
Changes in Short Physical Performance Battery (SPPB) from baseline | session 0 (initial visit); after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.
Changes in Four Square Step Test (FSST) from baseline | session 0 (initial visit); after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  FSST is used to assess dynamic stability and the ability of the subject to step over low objects forward, sideways, and backward.
Changes in EuroQol-5D (EQ-5D) from baseline | session 0 (initial visit); after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D questionnaire has two components: health state description and evaluation. In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are.
Changes in Fall Efficacy Scale-Korean (FES-K) from baseline | session 0 (initial visit); after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  FES-K is the measures of "fear of falling" or, more properly, "concerns about falling", which are suitable for use in research and clinical practice. A 10-item self-administered questionnaire designed to assess fear of falling in mainly community-dwelling older population.
Change in Muscle Strength from Baseline | session 0 (initial visit); after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  The maximal isometric strength of the 12 muscles in lower extremity will be measured with digital muscle testing device.
Change in Geriatric Depression Scale (GDS) from Baseline | session 0 (initial visit); after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  GDS is a 15-item self-report assessment used to identify depression in the elderly. A score of 0 to 5 is normal. A score greater than 5 suggests depression.
Change in 6 minute walk test (6MWT) from Baseline | session 0 (initial visit); after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
User Satisfaction Questionnaire | after session 12 (at approximately 4 weeks); after session 24 (at approximately 8 weeks)
  We evaluate the satisfaction questionnaire for GEMS-H use.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SH, Kim E, Kim J, Lee HJ, Kim YH. Robot-assisted exercise improves gait and physical function in older adults: a usability study. BMC Geriatr. 2025 Mar 22;25(1):192. doi: 10.1186/s12877-025-05811-1. PMID 40121407